CLINICAL TRIAL: NCT02375893
Title: The Official Title is in French: Microbiote, Acides Biliaires et Athérome Coronaire (MABAC)
Brief Title: Bile Acids and Gut Microbiota as Potent Coronary Atheroma Risk Factors: a Prospective Study in Human
Acronym: MABAC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A01643-44
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Coronary Disease
Keywords: Coronary disease; Bile acids; Gut microbiota; Risk factors; Atherosclerosis
MeSH Terms: conditions — Coronary Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Coronary patients: Feces, blood sample, clinical and biological data. Presence (1) of coronary disease defined as the presence of atheroma during the coronary angiogram
  Interventions: Other: No intervention
- Healthy subjects (2): Feces, blood sample, clinical and biological data. Absence (2) of atheroma during the coronary angiogram
  Interventions: Other: Healthy subject

INTERVENTIONS:
Other: No intervention — Collecting blood and feces samples
  Groups: Coronary patients
Other: Healthy subject — Collecting blood and feces samples
  Groups: Healthy subjects (2)

SUMMARY:
The purpose of this study is to describe the composition of bile acids and the gut microbiota comparing two populations: patients with coronary atheroma and the healthy subjects.

Our hypothesis is based on the demonstration of the anti atherogenic and anti inflammatory effect of certain bile acids, and the role of the gut microbiota in the metabolic regulation.

DETAILED DESCRIPTION:
Atherosclerosis is the main cause of cardiovascular diseases which remain the first cause of death worldwide. The prevention of risk factors can reduce the development of cardiovascular diseases. The final goal of our study is to find new protective or new risk factors that can be modulated to reduce the incidence of cardiovascular events.

Gut microbiota and its main metabolite, the bile acids, are implicated in the metabolic regulation. Some bile acids, especially the secondary bile acids, transformed from the primary bile acids by the bacteria of the gut microbiota, are now demonstrated in murine experimental atherosclerosis models, to be anti inflammatory and anti atherogenic molecules.

We want to compare the pool of bile acids and the composition of gut microbiota between the coronary patients and the healthy subjects to identify the potential protective or deleterious bacteria / bile acids.

All patients admitted for a scheduled coronary angiogram will be included, then divided into two groups: coronary or healthy, based on the presence or the absence of atheroma during the coronary angiogram.

Feces and blood samples, and clinical and biological data, will be collected during the patient's hospitalisation. No additional exam will be performed. The blood sample will be collected during the coronary angiogram or during a routine blood test.

ELIGIBILITY:
Inclusion Criteria:

- All patients admitted for a coronary angiogram

Exclusion Criteria:

* Statins, hypolipemic drugs, corticoids, anti HIV drugs
* Antibiotics adminisitration in the last 3 months
* Past of cholecystectomy
* Hepatic disorders
* Acute coronary syndrome
* No agreement, Insufficiency in comprehension
* Non fasting for at least 8 hours

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care center: cardiology unit.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition in coronary patients versus healthy subject | 8 months
  Observational only

SECONDARY OUTCOMES:
Bile acids composition in coronary patients versus healthy subjects, in feces and blood samples | 8 months
  Observational

CONTACTS AND LOCATIONS:
Overall Officials: Denis Duboc, MD, PhD, Principal Investigator — APHP
Locations (1):
- Cardiology Department, Cochin Hospital, Paris, France

REFERENCES:
- [Result] Chong Nguyen C, Duboc D, Rainteau D, Sokol H, Humbert L, Seksik P, Bellino A, Abdoul H, Bouazza N, Treluyer JM, Saadi M, Wahbi K, Soliman H, Coffin B, Bado A, Le Gall M, Varenne O, Duboc H. Circulating bile acids concentration is predictive of coronary artery disease in human. Sci Rep. 2021 Nov 22;11(1):22661. doi: 10.1038/s41598-021-02144-y. PMID 34811445